CLINICAL TRIAL: NCT06406530
Title: Topical Application of PRF in Tooth Extraction Sockets Before Radiation Therapy for Head and Neck Cancer
Brief Title: Topical Application of PRF Before Radiation Therapy
Acronym: PRF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Sameh Attia, Senior Physician in the department of Oral and Maxillofacial Surgery,PD, Dr. med. dent., M.Sc., University of Giessen
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TAPRFPR
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: PRF
Keywords: PRF; wound healing; dentistry; oral surgery; radiation therapy; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator
Masking Description: Investigator as well as the Patient are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRF site (test site) (Experimental): The participants become at least two teeth removed, one site is applied with PRF (test site) while the other is left for natural healing by forming a blood clot (control site). Operator and Investigator as well as the Patient are blinded to to the site of application.
  Interventions: Procedure: PRF
- Blood clot (control site) (Active Comparator): The participants become at least two teeth removed, one site is applied with PRF (test site) while the other is left for natural healing by forming a blood clot (control site). Operator and Investigator as well as the Patient are blinded to to the site of application.
  Interventions: Procedure: Natural Healing

INTERVENTIONS:
Procedure: PRF — Patients blood is standardized centrifuged and split in to a red-phase (erythrocytes) and white-phase (PRF). The gained PRF is processed to a clot-fort and is inserted into the alveolus.
  Other Names: Platelet rich fibrin
  Arms: PRF site (test site)
Procedure: Natural Healing — After the tooth extraction, natural healing is aimed by allowing a blood clot formation without any further intervention.
  Other Names: Blood clot formation
  Arms: Blood clot (control site)

SUMMARY:
The primary goal of this study is to observe whether PRP promotes the wound healing before a radiation therapy or not, compared to the natural healing of a tooth extraction socket.

Secondary aim is to monitore the effect on the pain perception.

DETAILED DESCRIPTION:
Head and neck cancer patients are required for a dental checkup before the beginning of the radiation therapy. During this checkup the patients gets a radiological and clinical examination in order to determine any tooth or alveolar bone bound inflammatory processes. Teeth associated to those conditions, or those which are likely to result in any of this, have to be extracted in order to prevent radiation associated complications such as osteomyelitis or further osteoradionecrosis of the jaw. In order to prevent this illness it is essential to not start before the healing of the post-extraction socket has reached a sufficient state, which is usually around 3 weeks post-extracitonem. To facilitate the healing, recent studies have shown an positive effect by applying PRF and a lower pain perception after surgical tooth removal. So far it is not documented for the prevention of a osteoradionecrosis of the jaw.

The patients who receive two or more tooth extractions before radiation therapy can participate in the study. The preliminary diagnosis has to be a head and neck tumor which is planned to be treated with ionizing radiation equally on both sides of the jaw(s). Both teeth have to have a similar size (e.g. molar and molar).

Patient and Doctors a blinded, the site of PRF Application is chosen by random. After surgical removal of the teeth one extraction socket is filled with PRF while the other is left for its natural formation of a blood clot.

During the first 7 days the patient protocols the pain perception and the amount of painkillers used for both sides of the jaw. After 7d, 14d, 21d, 30d, the wound healing is recorded until it reached is end in complete epithelization.

3 Months after the surgery a intermediate clinical examination is performed for early signs of any complication due to the radiation therapy. 6 Months after the surgery a OPG-radiograph will be taken to determine the bone healing comparing the test site and the control site.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer with planed radiation therapy
* Bilateral tooth extraction
* Similar tooth size
* Atraumatic tooth extractions without flap surgery
* Patients age above 18y of age

Exclusion Criteria:

* Prior radiation therapy in the head and neck area
* Prior and current therapy with bisphosphonates or equivalent modern biologics
* Patients during pregnancy or breastfeeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Wound healing between the two sites using the Wound Healing Index | around 4 Weeks
  To compare the wound heeling, a modified Landry and Turnbull Healing Index is used. This index varies from 0 to 5, where 0 means no healing and 5 excellent healing.

SECONDARY OUTCOMES:
PRF and Pain perception | around 7 days
  To compare pain perception between the two sites - the PRF test site and the control site - a visual analogue scale (VAS) for pain is provided to the patients. This scale ranges from 0 to 10, where 0 indicates no pain and 10 represents the highest imaginable pain for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Attia, DDS, MSc, Study Director — UKGM
Locations (1):
- University of Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided